CLINICAL TRIAL: NCT00607815
Title: A Comparison of CPT vs PCT for Veterans
Brief Title: A Comparison of Cognitive Processing Therapy (CPT) Versus Present Centered Therapy (PCT) for Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MHBA-007-07F
Record Dates: First submitted 2008-02-04; First posted 2008-02-06 (Estimated); Results first posted 2015-07-20 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-03

CONDITIONS: PTSD
Keywords: PTSD; OEF/OIF; Combat; Treatment; CPT; PCT; Cognitive
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Processing Therapy (Active Comparator): Cognitive Processing Therapy
  Interventions: Behavioral: Cognitive Processing Therapy
- Present Centered Therapy (Active Comparator): Present Centered Therapy
  Interventions: Behavioral: Present Centered Therapy

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — CPT is a highly structured protocol in which the client learns the skill of recognizing and challenging dysfunctional cognitions, first about the worst traumatic event and then later with regard to the meaning of the events for current beliefs about self and others.
  Arms: Cognitive Processing Therapy
Behavioral: Present Centered Therapy — Present centered therapy is a supportive counseling model developed by Drs. Foa and Shea. The treatment is called "present centered therapy" to 1) emphasize the need to focus on the participant's current life and 2) to conceptualize the problems as being caused by PTSD, and in some cases they may have been present for a long period of time. The treatment makes a connection between PTSD and current problems thus making it a more realistic PTSD treatment and still allowing PCT to control for nonspecific therapeutic factors
  Arms: Present Centered Therapy

SUMMARY:
The purpose of this study is to compare the effectiveness of Cognitive Processing Therapy (CPT) versus Present Centered Therapy (PCT) for male OEF/OIF Veterans with combat related PTSD.

DETAILED DESCRIPTION:
The purpose of this study is to compare the effectiveness of Cognitive Processing Therapy (CPT) versus Present Centered Therapy (PCT) for male OEF/OIF Veterans with combat related PTSD.

CPT has been shown to be effective in treating trauma survivors in several treatment outcome studies, but utility with Veterans has only been examined with male Veterans in one small pilot study. In addition CPT has never been compared to a treatment as usual or supportive psychotherapy condition to control for the specific and nonspecific elements of treatment. Although Cognitive Processing Therapy is one of the main treatment modalities at several VA's, including Cincinnati, it has never been compared to PCT, nor has it been used in a large, randomized study of male OEF/OIF Veterans. It is hypothesized that individual receiving CPT will show a larger reduction in posttraumatic stress disorder and related symptoms than those individuals receiving PCT.

All male OEF/OIF Veterans will be screened for their appropriateness for the study by phone screen and then by an assessment technician. The Veteran will be assessed at pre, post, 3-month, and 1-year follow-up. The assessment technicians will be blind to the participant's condition. CPT is a 12 week long individual psychotherapy treatment shown to be effective at reducing PTSD and related symptoms for survivors of various types of traumas, including combat. PCT is a supportive counseling treatment that has been utilized as an alternative to waitlist control in VA cooperative studies of PTSD.

ELIGIBILITY:
Inclusion Criteria:

* PTSD;
* memory of the trauma;
* able to read/write;
* must be stable on medication for 3 months

Exclusion Criteria:

* Psychosis;
* suicidal/homicidal intent;
* alcohol/substance dependence;
* no memory of the trauma

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must be a male combat Veteran
Enrollment: 79 (Actual)
Dates: Start 2009-06-15 (Actual); Primary Completion 2015-02-01 (Actual); Study Completion 2015-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Chard, PhD, Principal Investigator — Cincinnati VA Medical Center, Cincinnati, OH
Locations (1):
- Cincinnati VA Medical Center, Cincinnati, OH, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Processing Therapy | Present Centered Therapy
Started | 43 | 36
Completed | 20 | 25
Not Completed | 23 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Processing Therapy | Present Centered Therapy | Total
Number analyzed (Participants) | 43 | 36 | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (7.11) | 32.11 (7.85) | 30.92 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 43 | 36 | 79
Clinician Administered PTSD Scale [Mean (Standard Deviation); unit: units on a scale] — Clinician-rated PTSD symptom severity; higher is worse; range at post-treatment is 0 to 80; scale scores are summed.
  units on a scale | 60.14 (11.61) | 62.42 (14.84) | 61.77 (13.14)
PTSD Checklist [Mean (Standard Deviation); unit: units on a scale] — 17-item patient self-reported PTSD severity; higher is worse; range at post-treatment is 17-73; scale scores are summed.
  units on a scale | 53.83 (9.87) | 53.49 (9.33) | 53.65 (9.52)
Beck Depression Inventory [Mean (Standard Deviation); unit: units on a scale] — Gold-standard, self-reported depression severity measure; higher is worse; post-treatment range is 2-45. scale scores are summed.
  units on a scale | 27.70 (9.68) | 28.22 (10.21) | 27.94 (9.86)
State Trait Anxiety [Mean (Standard Deviation); unit: units on a scale] — Self-reported trait anger; subscale score is summed; higher is worse; range at post-treatment is 10-37.
  units on a scale | 43.19 (5.60) | 43.14 (4.18) | 43.17 (4.84)
State Trait Anger Expression Inventory [Mean (Standard Deviation); unit: units on a scale] — Self-reported state anxiety; higher is worse; scale score is summed; range at post-treatment is 20-73.
  units on a scale | 28.14 (5.52) | 26.35 (6.07) | 27.16 (5.86)

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale
Description: Clinician-rated PTSD symptom severity; higher is worse; range at post-treatment is 0 to 80; scale scores are summed.
Time Frame: Post-treatment, at 3 months and 1 year
Population: Generalized estimating equations (GEE) were used to test study hypotheses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Processing Therapy | Present Centered Therapy
Number analyzed (Participants) | 43 | 36
units on a scale
  post | 31.56 (21.24) | 42.62 (23.76)
  3-month | 31.65 (21.77) | 38.73 (18.38)
  12-month | 26.78 (19.26) | 32.12 (22.48)

2. Primary Outcome: PTSD Checklist (PCL)
Description: 17-item patient self-reported PTSD severity; higher is worse; range at post-treatment is 17-73; scale scores are summed
Time Frame: post-treatment, at 3 months and 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Processing Therapy | Present Centered Therapy
Number analyzed (Participants) | 43 | 36
units on a scale
  post | 33.48 (15.75) | 42.88 (23.76)
  3-month | 35.55 (14.17) | 41.84 (14.66)
  12-month | 33.72 (13.69) | 34.88 (12.32)

3. Secondary Outcome: Beck Depression Inventory - II (BDI-II)
Description: Gold-standard, self-reported depression severity measure; higher is worse; post-treatment range is 2-45. scale scores are summed.
Time Frame: post-treatment, at 3 months and 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Processing Therapy | Present Centered Therapy
Number analyzed (Participants) | 43 | 36
units on a scale
  post | 16.32 (11.42) | 20.73 (10.53)
  3-month | 17.10 (10.48) | 18.95 (9.67)
  12-month | 15.56 (12.41) | 18.47 (11.96)

4. Secondary Outcome: State-Trait Anger Scale (STAXI)
Description: Self-reported trait anger; subscale score is summed; higher is worse; range at post-treatment is 10-37.
Time Frame: post-treatment, at 3 months and 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Processing Therapy | Present Centered Therapy
Number analyzed (Participants) | 43 | 36
units on a scale
  post | 21.75 (5.58) | 23.81 (6.69)
  3-month | 21.26 (6.49) | 23.09 (5.04)
  12-month | 21.64 (7.09) | 22.41 (3.95)

5. Secondary Outcome: State-Trait Anxiety Scale
Description: Self-reported state anxiety; higher is worse; scale score is summed; range at post-treatment is 20-73.
Time Frame: post-treatment, at 3 months and 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Processing Therapy | Present Centered Therapy
Number analyzed (Participants) | 43 | 36
units on a scale
  post | 43.20 (13.71) | 48.34 (11.42)
  3-month | 44.98 (12.92) | 47.21 (13.20)
  12-month | 43.27 (13.39) | 45.71 (12.29)

ADVERSE EVENTS:
Arm/Group | Cognitive Processing Therapy | Present Centered Therapy
Serious Adverse Events (participants affected / at risk) | 1/43 | 0/36
Other Adverse Events (participants affected / at risk) | 0/43 | 0/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Processing Therapy (N=43) | Present Centered Therapy (N=36)
Self Harm (Psychiatric disorders) | 1 (1) | 0 (0) — Pt had a fight with mother over his recent relapse to substances. Pt was admitted for passive self-harm thoughts. Pt completed 8 sessions of therapy with a significant reduction in PTSD symptoms. The event was found to be unrelated by the IRB.

LIMITATIONS AND CAVEATS:
Significant amounts of missing data from patients not attending assessment. Drop out rate from treatment was higher than other clinical trials of CPT and PCT in civilian samples, but in keeping with other studies of Veterans.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes